CLINICAL TRIAL: NCT02738593
Title: Using Next Generation Sequencing (NGS) Method to Detect Circulating Free DNA (Cf-DNA) and Explore the Resistance and Prognosic Mechanism of Third Generation Epidermal Growth Factor Receptor (EGFR) Tyrosine-kinase Inhibitor (TKI) in Advanced Non-small Cell Lung Cancer (NSCLC) Patients: a Single Center Study
Brief Title: Detection Cell Free DNA in Lung Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Li Zhang, Profressor, Sun Yat-sen University
Other Study IDs: TKI0301
Record Dates: First submitted 2016-04-06; First posted 2016-04-14 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — periphereal blood 10ml,centrifuge:4℃、2400g、10min,extracted plasma and stored in -80° refrigerator.
  fresh tumor tissue sample,store in freezing medium within 2 hours. FFPE tumor tissue.
Oversight: Data Monitoring Committee: No

SUMMARY:
third generation of EGFR-TKIs is the newest target therapy for NSCLC. However, we did not known the specific mechanisms for those non-responders and patients grow resistance.Next generation sequencing is current the most sensitive and specific method to exam gene mutation, diversion etc.

By consistently detect the cf-DNA, we could possibly find out the mechanisms of response and resistance.

DETAILED DESCRIPTION:
Study backgroud: third generation of epidermal growth factor receptor tyrosine kinase inhibitors (EGFR-TKIs) is the newest target therapy for non small cell lung cancer (NSCLC). Two major study published in NEJM show that the overall response rate is about 60%-70%, with a progression free survival about 10 months. However, we did not known the specific mechanisms for those non-responders and patients grow resistance.

Next generation sequencing is current the most sensitive and specific method to exam gene mutation, diversion etc. By consistently detect the cf-DNA, we could possibly find out the mechanisms of response and resistance.

Eligible patients received 3rd generation EGFR-TKIs (AZD9291 and AVITINIB) were enrolled into this study. Tumor tissue sample within 6 months, and 10ml periphereal blood samples were collected at baseline. After treatment initiation, 10ml periphereal blood would be collected at every image testing time point until disease progression. Blood samples will be draw using EDTA tube and centerfuged within 2 hours and store in -80 refrigerator.

NGS testing will cover target genes of NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* pathologically confirmed non small cell lung cancer.
* harboured with positive EGFR mutation (19 exon deletion, L858R、G719X、L861Q mutation)
* reliable patients history data.

Exclusion Criteria:

* pathologically not confirmed non small cell lung cancer.
* multiple primary cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced non-small cell lung cancer (NSCLC),prepare to receive third generation of epidermal growth factor receptor tyrosine kinase inhibitors (EGFR-TKIs) treatment. Patients must harboured with positive EGFR mutation (19 exon deletion, L858R、G719X、L861Q mutation), able to provide periphereal blood and tumor tissue.
Sampling Method: Non-Probability Sample
Enrollment: 124 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-04 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
cf-DNA change from baseline | baseline and every 2 months up to 36 months or first documented progression disease.
  Using next generation sequencing (NGS) method to detect circulating free DNA (cf-DNA) in patients receive third generation EGFR-TKI, periphereal blood sample were collected at baseline and every 2 months to disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, Principal Investigator — Sun Yat-sen University
Locations (2):
- China (2):
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: Undecided